CLINICAL TRIAL: NCT01986218
Title: Phase I Ascending Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-986115 in Subjects With Advanced Solid Tumors
Brief Title: Phase I Ascending Multiple-Dose Study of BMS-986115 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: (Non-safety reason, business objectives have changed)
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA002-001
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Various Advanced Cancer
MeSH Terms: interventions — BMS-986115

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A: Dose Escalation (BMS-986115) (Experimental): Continuous daily dosing until disease progression or unacceptable toxicity
  Interventions: Drug: BMS-986115
- Arm A: Dose Expansion (BMS-986115) (Experimental): Continuous daily dosing until disease progression or unacceptable toxicity
  Interventions: Drug: BMS-986115
- Arm B: Dose Escalation (BMS-986115) (Experimental): Twice weekly dosing until disease progression or unacceptable toxicity
  Interventions: Drug: BMS-986115
- Arm B: Dose Expansion (BMS-986115) (Experimental): Twice weekly dosing until disease progression or unacceptable toxicity
  Interventions: Drug: BMS-986115

INTERVENTIONS:
Drug: BMS-986115
  Other Names: BMS-986115 (Notch Inhibitor)

SUMMARY:
The primary purpose of this study is to evaluate the safety and effectiveness of daily doses of BMS-986115 in subjects with advanced solid tumors

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Subjects with a histologically or cytologically confirmed diagnosis of solid tumors, advanced or metastatic, refractory to or relapsed from standard therapies or for which there is no known effective treatment
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1
* Prior anti-cancer treatments are permitted (i.e., chemotherapy, radiotherapy, hormonal, or immunotherapy)
* At least 4 weeks must have elapsed from last dose of prior anti-cancer therapy and the initiation of study therapy

Exclusion Criteria:

* Subjects with known or suspected brain metastases, primary brain tumors, or brain as the only site of disease
* Evidence of uncontrolled, active infection, requiring systemic anti-bacterial, anti-viral or anti-fungal therapy ≤ 7 days prior to administration of study medication
* Current or recent (within 3 months of study drug administration) gastrointestinal disease such as chronic or intermittent diarrhea, or disorders that increase the risk of diarrhea, such as inflammatory bowel disease. Non-chronic conditions (e.g. infectious diarrhea) that are completely resolved for at least 2 weeks prior to starting study treatment are not exclusionary
* Any major surgery or gastrointestinal disease that would interfere with administration of oral medications
* Conditions requiring chronic systemic glucocorticoid use, such as autoimmune disease or severe asthma, excluding inhalation steroids for maintenance.
* Uncontrolled or significant cardiovascular disease
* History of medically significant thromboembolic events or bleeding diathesis within the past 6 months
* Inadequate bone marrow function (Absolute neutrophil count (ANC) < 1,500 cells/mm3; Platelet count < 100,000 cells/mm3; Hemoglobin < 9.0 g/dL)
* Inadequate hepatic function (Total bilirubin > 1.5 times the institutional upper limit of normal (ULN) (except known Gilbert's syndrome); Alanine transaminase (ALT) or aspartate transaminase (AST) > 2.5 times the institutional ULN. ALT or AST up to 3 times the institutional ULN permitted if total bilirubin is normal
* Uncontrolled (≥ Grade 2) hypertriglyceridemia (fasting triglycerides > 300 mg/dL (3.42 mmol/L))
* Inadequate renal function (Blood creatinine > 1.5 times the institutional ULN)
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or Human Immunodeficiency Virus (HIV) -1, -2 antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple daily doses of BMS-986115 | Up to 30 days after the last dose of study medication (approximately 18 months)
  Measured by the frequency of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, Grade 3 or 4 AEs, deaths, laboratory abnormalities and clinically relevant electrocardiogram (ECG) changes from baseline

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986115 and its active metabolite BMT-100948 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Time of maximum observed plasma concentration (Tmax) of BMS-986115 and its active metabolite BMT-100948 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Trough observed plasma concentration (Ctrough) of BMS-986115 and its active metabolite BMT-100948 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of BMS-986115 and its active metabolite BMT-100948 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-986115 and its active metabolite BMT-100948 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Area under the concentration-time curve in one dosing interval [AUC(TAU)] of BMS-986115 and its active metabolite BMT-100948 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Terminal plasma half-life (T-HALF) of BMS-986115 and its active metabolite BMT-100948 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Apparent total body clearance (CLT/F) of BMS-986115 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Apparent volume of distribution at steady-state (Vz/F) of BMS-986115 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
AUC Accumulation Index; ratio of AUC(TAU) at steady state to AUC(TAU) after the first dose (AI_AUC) of BMS-986115 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Ratio of metabolite AUC(INF) to parent AUC(INF) after single dose and ratio of metabolite AUC(TAU) to parent AUC(TAU) at steady state, corrected for molecular weight (MR_AUC) of BMS-986115 and its active metabolite BMT-100948 | 29 timepoints up to Cycle 3 Day 1 (approximately 32 days)
Pharmacodynamics (PD) changes in the expression of Notch pathway-related genes, including but not limited to Hes1 and Deltex1, as determined by standard molecular methods | 16 timepoints up to Cycle 2 Day 16 (approximately 20 days)
Preliminary anti-tumor activity of BMS-986115 as measured by response evaluation criteria in solid tumors (RECIST) | Screening (within 30 days prior to Day 1), Every 8 weeks, End of Treatment or 30-Day follow-up visits (approximately 18 months)
  Assessed by:
  * Tumor Response based on the Investigator's assessment using RECIST v1.1 [categorized as complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD)]
  * Best Overall Response (BOR), defined as the best tumor response recorded between the data of first dose and the last on-study tumor assessment (prior to any subsequent cancer therapy)
  * Overall Response Rate, defined as the proportion of subjects with BOR responses of CR or PR
  * Disease Control Rate, defined as the proportion of subjects with BOR responses of CR, PR or SD
  * Progression-Free Survival (or PFS), defined as time from first dose to either progressive disease, initiation of subsequent off-study therapy, or death

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Usc/Norris Comprehensive Cancer Center, Los Angeles, California, United States
- Local Institution, Parkville, Victoria, Australia
- Canada (2):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx